CLINICAL TRIAL: NCT02344212
Title: Weight Loss and Prevention in Latina Immigrants: Advancing Methods of Community-Based Intervention Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: UAB Diabetes Research Center (Unknown); UAB Nutrition Obesity Research Center (Unknown); UAB Minority Health & Research Center (Unknown); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: X080107001
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ESENCIAL Para Vivir (Experimental): Overweight or obese Latina immigrant women were recruited to participate an 8-week weight loss program to reduce or delay their risk of developing diabetes. Data was collected at baseline, program completion, and six months.
  Interventions: Behavioral: ESENCIAL Para Vivir: a weight loss program for Latinas

INTERVENTIONS:
Behavioral: ESENCIAL Para Vivir: a weight loss program for Latinas — Overweight or obese Latina immigrant women were recruited to participate an 8-week weight loss program to reduce or delay their risk of developing diabetes. Data was collected at baseline, program completion, and six months.
  Other Names: ESENCIAL Para Vivir; ESENCIAL: a weight loss program for Latina

SUMMARY:
The long-term objective of this study protocol is to develop and test a culturally sensitive, community-based intervention, ESENCIAL Para Vivir (Essential for Life) to promote weight loss and diabetes prevention among overweight or obese Latina immigrants. We chose to focus on Latinas because Latinas are at especially high risk for developing diabetes and currently there are not Spanish programs available in our area that provide education about weight management and diabetes prevention.

DETAILED DESCRIPTION:
The 8-week weight loss program, ESENCIAL Para Vivir (Essential for Life), is comprised of 6 groups sessions and 2 individual sessions delivered by a bilingiual, bi-cultural Community Health Advisor. All sessions are interactive with activities that build on educative content and most contain an interactive DVD component. We propose an innovative approach that will employ the DVD in tandem with our education sessions delivered by a Community Health Advisor to maximize buy-in from participants as well as provide access to community health leaders (medical professionals - endocrinologists, internists, nutritionists). Participants will be over 19 years of age, self-identifying as Hispanic women without diabetes, not pregnant or have given birth within the previous six months. The participants will be recruited from Jefferson County through community agencies and organization. Participants will be recruited and screened with an initial contact sheet to ensure that they meet our criteria, then they will be consented and complete baseline measurements. At the completion of the program, participants will repeat measures done at baseline, and 6 months post program completion.

ELIGIBILITY:
Inclusion Criteria:

* female aged 19 years or older,
* foreign born, self-identified as Latina,
* no history of diagnosed diabetes,
* fasting blood sugar < 126 mg/dL, and overweight or obese (BMI > 25kg/m2).

Exclusion Criteria:

* any medical condition for which weight loss was contraindicated; a fasting glucose > 126 mg/dL,
* pregnancy, postpartum less than 6 months, or planning a pregnancy before the end of the study period.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in weight | 6 months
  Change in weight from baseline to end of intervention (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Cherrington, MD MPH, Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Derived] Cherrington AL, Willig AL, Agne AA, Fowler MC, Dutton GR, Scarinci IC. Development of a theory-based, peer support intervention to promote weight loss among Latina immigrants. BMC Obes. 2015 Mar 19;2:17. doi: 10.1186/s40608-015-0047-3. eCollection 2015. PMID 26217532